CLINICAL TRIAL: NCT02579577
Title: Decision Making and Future Planning for Children With Complex Illnesses: a Qualitative Multi-stakeholder, Longitudinal Study.
Brief Title: Decision Making and Future Planning for Children With Complex Illness
Status: Completed | Type: Observational
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Other Study IDs: 15068
Record Dates: First submitted 2015-07-31; First posted 2015-10-19 (Estimated); Last update posted 2017-05-03 (Actual); Status verified 2016-05

CONDITIONS: Long-Term Care; Palliative Care
MeSH Terms: interventions — Observation; Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Decision making cohort: Any people identified as being important within the network of care for children with life-limiting illnesses.
  Interventions: Other: Observation; Other: Interviews; Other: Medical notes review

INTERVENTIONS:
Other: Observation — Observation of clinic appointments and ward rounds if the child is admitted to hospital during the study period.
Other: Interviews — Semi-structured interviews will be conducted approximately 3 times during the study period with each participant.
Other: Medical notes review — The child's electronic medical record will be accessed periodically to identify any planned appointments or periods of hospitalisation and their medical notes will also be reviewed at the end of the study.

SUMMARY:
The population of children with life-limiting illnesses (LLI) in England is increasing and there is growing need to improve the quality of children's palliative care. Families of children with LLI are confronted with many care decisions for their children, such as whether and when to commence artificial nutrition or ventilation. They may also have the opportunity to consider the care that may be appropriate for their child in the future. Despite the important decisions families and professionals are required to make, there is little empirical evidence regarding the process of decision making and future planning for this population. Few studies have investigated the perspectives of multiple stakeholders and none have addressed multiple perspectives longitudinally. Therefore the relational and contextual aspects of decision making and future planning for children with LLI have as yet not been identified.

A multiple embedded case study utilising ethnographic methods (semi-structured interviews, observation and notes review) is proposed to address this knowledge gap. Families of children with LLI cared for in either of two participating hospitals will be recruited and followed up for up to 12 months. The family will be invited to nominate 'significant others' (e.g. relatives, friends, health care professionals) who assist them in decision making and future planning, to participate in the study. Outpatient clinic appointments or ward rounds during periods of hospitalisation will be observed and semi-structured interviews will be conducted approximately three times with each participant. Medical notes will be reviewed at the end of the study.

This research will enable a better understanding of the experiences and preferences for engaging in decision making and future planning from the perspectives of all stakeholders. It will also provide an awareness of the communication practices involved in discussions and the networks of care surrounding children with LLI, including specific support needs in relation to their role.

ELIGIBILITY:
Inclusion criteria - Parent

* Their child must be between 28 days and 18 years old
* Their child must have a LLI within categories 2-4 (Association for Children with Life-threatening and Terminal Conditions and their Families, 2004) (see page 8)
* Child must be under the care of a consultant at either of the two NHS Trusts included in the study
* The parent must be aware of the child's LLI diagnosis
* Participants must speak English. This is both due to resource constraints and due to the sensitive topic such that difficulties in translating questions sensitively may cause greater distress to participants.

Inclusion criteria - Child

* Children will be classed as participants if their parent is a participant and consents to their child's medical notes being accessed.
* For children to participate in the interview component of the study, they must be over the age of 7 years and cognitively able to provide their own assent (or consent, if over 16 years old)
* Parents must have agreed to the child's participation if they are under 16 years old
* Participants must speak English or be able to communicate in some way using alternative or augmentative communication.

Inclusion criteria - Significant Others/Professionals

* Significant others must have been identified by the eligible child and/or parents as being important in their decision making and future planning
* Participants must speak English
* Participants must be over the age of 7 years and provide their own assent alongside parental consent (if under 16 years old) or provide consent if they are over the age of 16 years (in the case of a friend or sibling being nominated as a 'significant other').

Exclusion Criteria:

* Families and significant others of children with ACT Category 1 life-threatening illnesses (Conditions for which curative treatment may be feasible but can fail)
* Participants who do not meet the inclusion criteria.

Min Age: 28 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Each case will be centred around a child with a life-limiting illness and their parents who will have been identified as eligible by their usual care team. Additional significant others who are important in their decision making and future planning will be identified by the family and will ideally include at least one health professional. However, the composition of each case will be determined by the child and family and may involve only them. Nominated 'significant others' may include extended family, peers, ministers of religion, key workers etc.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2015-10; Primary Completion 2017-01-31 (Actual); Study Completion 2017-01-31 (Actual)

PRIMARY OUTCOMES:
Semi-Structured Interview Responses | Up to 24 months
  Interviews will be semi-structured, with a broad opening question asking the participant about the child at the centre of the case; both in terms of their illness and their context (family, personality, values and goals). Although the topics of decision making and future planning will be covered within the interview, the way in which these are initiated are likely to be different for each participant and asked in relation to the responses given to the opening question.
Observational fieldnotes | Up to 24 months
  Observations will occur at clinic appointments and ward rounds and will aim to identify the communication processes involved in decision making and how each individual involved participates.

CONTACTS AND LOCATIONS:
Overall Officials: Bridget Johnston, Professor, Principal Investigator — University of Nottingham
Locations (3):
- United Kingdom (3):
  - Sherwood Forest Hospitals NHS Trust, Mansfield
  - Nottingham University Hospitals NHS Trust, Nottingham
  - Sheffield Children's Hospital, Sheffield